CLINICAL TRIAL: NCT06578429
Title: Deep TMS Neuromodulation of Neural Circuits Associated With Stimulant Use Disorder
Brief Title: Deep TMS of Neural Circuits Associated With Stimulant Use Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: VA Palo Alto Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Claudia Padula, Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 72401
Record Dates: First submitted 2024-08-26; First posted 2024-08-29 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Methamphetamine Use Disorder; Transcranial Magnetic Stimulation
Keywords: Veterans; Deep Transcranial Magnetic Stimulation (dTMS); Neuroimaging; Relapse
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, sham-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization will be completed and stored with staff in the Biostatistic Core. Treatment assignments will be recorded on a USB drive read by the device in order to ensure treaters and study investigators remain blinded. In the instance that a serious adverse event (SAE) occur, consultation with the Data Safety and Monitoring Board and the Institutional Review Board will occur to determine the appropriateness of breaking the blind. The blind may be broken for a specific individual in order to determine whether the SAE is related to the treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active dTMS (Experimental): Participants will receive 30 active dTMS treatments, administered 3 times per day over 10 consecutive business days. Each treatment visit will last approximately 30 minutes in total.
  Interventions: Device: Deep Transcranial Magnetic Stimulation (dTMS) H4 coil - Active
- Sham dTMS (Sham Comparator): Participants will receive 30 sham dTMS sessions, administered 3 times per day over 10 consecutive business days. Each treatment visit will last approximately 30 minutes in total.
  Interventions: Device: Deep Transcranial Magnetic Stimulation (dTMS) H4 coil - Sham

INTERVENTIONS:
Device: Deep Transcranial Magnetic Stimulation (dTMS) H4 coil - Active — The study will utilize the H4 coil to administer active Deep Transcranial Magnetic Stimulation (dTMS) to the bilateral insula, a core salience network node.
  Arms: Active dTMS
Device: Deep Transcranial Magnetic Stimulation (dTMS) H4 coil - Sham — The study will utilize an identical protocol using the H4 coil to administer a sham condition.
  Arms: Sham dTMS

SUMMARY:
This study aims to evaluate the efficacy of deep transcranial magnetic stimulation (dTMS) as a treatment for Veterans with a methamphetamine use disorder (MUD).

DETAILED DESCRIPTION:
To date, TMS has emerged as a promising treatment avenue for addiction and is being tested in clinical trials with some encouraging results. A recent systematic review and meta-analysis highlights that 7/8 (87.5%) studies using TMS for MUD or 38/50 (88%) in addiction more broadly have targeted the left DLPFC alone. While this strategy has been useful in reducing craving, treated individuals resume use shortly after treatment at similar rates to those receiving sham. Here, utilizing a data-driven and innovative approach, the investigators aim to modulate target brain function that has been shown to predict treatment outcomes for individuals with MUD. The literature describes how TMS treatment is associated with physiological changes in the brain at the target area and in remote structurally or functionally connected brain areas. TMS has been associated with changes in long-term potentiation (LTP) or depression (LTD) to increase neuroplasticity through increases in brain-derived neurotrophic factor (BDNF) and implicated in influencing the excitatory/inhibitory balance of GABAergic synapses. H-coil designs have the potential to target deeper regions of the brain as well as multiple downstream, interacting brain networks in a novel manner. For example, insula stimulation has the potential to strengthen the salience network broadly and subsequently ameliorate relapse risk.

An emerging advancement is the use of coils that target deeper regions of the brain and have the potential of targeting multiple, interacting brain networks. The H-coil configuration in this technique stimulates a broader area (e.g., up to 17 cubic centimeters) as well as a deeper area (e.g., up to 4 cm), relative to standard figure-of-eight coils, further enhancing innovation and generalizability. With this coil, the investigators hypothesize modifying the salience network nodes that are otherwise not reached by figure-of-eight coils. Notably, published studies to date that utilize these H-coils for addiction yield promising results. However, whether the proposed stimulation strategies will have objectively measurable impact on their respective brain targets or similar impact in individuals with MUD remains unclear.

The proposed study fills a critical, scientific gap of the need to evaluate a novel, non-invasive brain stimulation technique for MUD.

The investigators believe this proposed work will provide preliminary data for a larger grant submission that could allow for a more complex study design to fully answer gaps in current knowledge about deep TMS H4 coil as a possible treatment approach for MUD.

ELIGIBILITY:
Inclusion:

* Must be within the age range of 25-75.
* Participants must meet Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria for moderate to severe MUD (≥4 diagnostic symptoms).
* Participants must be able to obtain a Motor Threshold (MT), which will be determined during the screening process.
* Participants must have an adequately stable condition and environment to enable attendance at scheduled clinic visits.
* Participants must be able to read, verbalize, understand, and voluntarily sign the Informed Consent Form prior to participation in study procedures in English.
* If participants are on a medication regimen for comorbid symptoms, that regimen will be stable for the duration of the study and patient will be willing to remain on this regimen during the treatment phase.
* Participants must be fluent in English

Exclusion criteria:

* Transcranial magnetic stimulation (TMS) and magnetic resonance imaging (MRI) contraindications: such as a cardiac pacemaker, cochlear implant, or an implanted device (deep brain stimulation, ferromagnetic metal in the head and body, claustrophobia, pregnant or breastfeeding or other ferromagnetic device/object in the head and body within 30 cm of the treatment coil.
* General medical condition, disease, or neurological disorder that interferes with the assessments or participation.
* Unable to safely withdraw, at least two weeks prior to treatment, from medications that increase seizure risk.
* Current substance abuse as determined by positive toxicology screen
* Have a mass lesion, cerebral infarct, or other active CNS disease, including a seizure disorder.
* A recent suicide attempt (defined as within the last 30 days) or presence of current suicidal plan or intent. Patients at risk for suicide will be required to establish a written safety plan involving their primary therapist before entering the study.
* Severe impediment to vision, hearing and/or hand movement, as this is likely to interfere with the ability to follow study protocols.
* Greater than mild traumatic brain injury (defined as greater than 10 minutes loss of consciousness).
* Taking benzodiazepines or neuroleptic medications, or any medication known to alter seizure threshold.
* Acute or unstable chronic illness.
* Current or lifetime history of bipolar disorder or psychosis.
* Participation in another concurrent intervention-based clinical trial.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Insula Function | 1-4 days post-treatment
  The primary measure of SN function will include insula activation during the monetary incentive delay task, anticipation of loss contrasted with no loss
Percentage of Days Abstinent | 3 months post-treatment
  Methamphetamine use outcomes will be assessed using the TimeLine Follow Back (TLFB) Method, which utilizes calendar cue to recall recent, self-reported substance use, combined with objective biomarker data

SECONDARY OUTCOMES:
Other Salience Network Function | 1-4 days post-treatment
  The secondary measures of SN function will include insula to PFC functional connectivity, and dACC to insula functional connectivity using the same task as the primary measure.
Resting-State Salience Network | 1-4 days post-treatment
  The investigators will also utilize whole-brain, voxel-wise analyses for the task with stringent error correction, as well as insula activation and insula to dACC functional connectivity during resting state fMRI.
Binary Relapse | 3 months post-treatment
  Binary (yes/no) relapse after treatment via self-report

CONTACTS AND LOCATIONS:
Overall Officials: Claudia B Padula, PhD, Principal Investigator — Stanford University; Michelle R Madore, PhD, Principal Investigator — Stanford University
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Any data, specimens, forms, reports, and other records that leave the site will be identified only by a participant ID number to maintain confidentiality. The ID Number will have no relationship to any aspect of identifiable private information. Therefore, the data associated with each participant will be completely de-identified and there will be no mechanism by which users can re-identify participant data (e.g., name, address) with the subject code.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Three to twelve months after publication.
Access Criteria: Researchers who provide a methodologically sound proposal.

REFERENCES:
- [Background] Koob GF, Volkow ND. Neurocircuitry of addiction. Neuropsychopharmacology. 2010 Jan;35(1):217-38. doi: 10.1038/npp.2009.110. PMID 19710631
- [Background] Peters SK, Dunlop K, Downar J. Cortico-Striatal-Thalamic Loop Circuits of the Salience Network: A Central Pathway in Psychiatric Disease and Treatment. Front Syst Neurosci. 2016 Dec 27;10:104. doi: 10.3389/fnsys.2016.00104. eCollection 2016. PMID 28082874
- [Background] Harel M, Perini I, Kampe R, Alyagon U, Shalev H, Besser I, Sommer WH, Heilig M, Zangen A. Repetitive Transcranial Magnetic Stimulation in Alcohol Dependence: A Randomized, Double-Blind, Sham-Controlled Proof-of-Concept Trial Targeting the Medial Prefrontal and Anterior Cingulate Cortices. Biol Psychiatry. 2022 Jun 15;91(12):1061-1069. doi: 10.1016/j.biopsych.2021.11.020. Epub 2021 Dec 6. PMID 35067356
- [Background] Gay A, Cabe J, De Chazeron I, Lambert C, Defour M, Bhoowabul V, Charpeaud T, Tremey A, Llorca PM, Pereira B, Brousse G. Repetitive Transcranial Magnetic Stimulation (rTMS) as a Promising Treatment for Craving in Stimulant Drugs and Behavioral Addiction: A Meta-Analysis. J Clin Med. 2022 Jan 26;11(3):624. doi: 10.3390/jcm11030624. PMID 35160085